CLINICAL TRIAL: NCT00447174
Title: Dyadic Therapy Assessment Among Couples Coping With Traumatic Loss of a Child
Brief Title: Parental Bereavement Study Among Couples Coping Traumatic Loss of a Child
Acronym: PBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herzog Hospital (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BromD1CTIL
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Bereaved Parents
Keywords: Grief; parental bereavement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment (Experimental): treatment manual
  Interventions: Behavioral: Dyadic treatment for parental bereavement
- control group (No Intervention)

INTERVENTIONS:
Behavioral: Dyadic treatment for parental bereavement
  Arms: treatment

SUMMARY:
1. Develop a treatment for clinically significant parental bereavement. The proposed treatment development activities include:

   1. Development of a treatment manual, associated fidelity rating forms, and training aids,
   2. Pre-testing the treatment manual with bereaved parents, and revision in consultation with treatment development experts,
2. Conduct a randomized, wait-list control, pilot study of the proposed treatment:

   1. Measure treatment-related change in (a) complicated grief symptoms, the primary outcome variable, which will be assessed using the Inventory of Complicated Grief, and, (b) marital adjustment, the secondary outcome measure, to be assessed using the Dyadic Adjustment Scale. These outcomes will be assessed in treatment and control groups at baseline, at treatment conclusion, and at three month follow-up.
   2. Test the difference between the treatment and control groups on changes from baseline to three month follow-up on the exploratory outcome variables of PTSD, depression, social and work impairment, and quality of life
   3. Estimate effect sizes of these differences in changes in outcomes
3. Develop a proposal for a randomized controlled trial of the treatment, based on the results of aim 2.

DETAILED DESCRIPTION:
RESEARCH DESIGN AND METHODS

Treatment Manual Development: Psychoeducation, Dyadic Communication in Adversity, Stress inoculation training and skills building, Cognitive processing and restructuring, Exposure through constructive narrative.Reconstruction of a positive future and relapse prevention..

WAIT-LIST CONTROL STUDY Once the treatment manual is developed, we will move immediately into pilot testing of the treatment in bereaved families. The design for this pilot study is repeated measures that compares two groups at three time points of assessment: (pre-treatment, immediately post-treatment, 3 months post-treatment). Although other outcomes will be assessed, the primary outcomes will be a measure of bereavement and a measure of marital adjustment. The three month follow-up results will be compared to the pre-treatment results using an intent-to-treat analysis with the last observation carried forward. As treatment can last from 13 to 16 sessions, the wait-list control group's welfare is of concern. We will use weekly phone conversations to check in with wait-list participants. If they appear to be deteriorating, they will be immediately referred for treatment. Wait-list participants will be offered treatment at the end of the wait-list period. It should be noted that this contact during the wait-list period represents attention provided to wait-list participants, and thus makes our design somewhat conservative. It is the primary purpose of this study to establish preliminary efficacy through investigating effect sizes associated with the treatment, and to develop a treatment manual, and other required tools to conduct a full efficacy trial.

Participants. Participants will be parents living in Israel who have lost a child, are at least 6 months post loss (following Shear), are over the age of 21, can provide informed consent, and score > 30 on the Inventory of Complicated Grief. Subjects meeting these criteria will undergo a structured clinical interview to assess for inclusion and exclusion criteria. Participants will be provided free treatment, and if needed because of income restrictions will be provided with aid to defray transportation costs to the clinic.

Subject Recruitment. We will be using various methods of recruitment, including press as well as working with partnering organizations who deal with parental bereavement , and recruitment through the trained therapists who work in different clinical settings.

Assessor Training. Assessors will be trained on all measures They are psychometric measures and will be used as specified in the manuals that pertain to their use.

Independent Assessment. Assessors will be kept unaware of what treatment condition the person is in.

Demographics and Bereavement History. In addition to standard demographic information, we will obtain detailed information about the circumstances surrounding the child's death .

Psychiatric History. Axis I disorders will be assessed using the Structured Clinical Interview for DSM-III-R (SCID-1).The SCID is a semi-structured interview commonly used in research settings to assess a subject's psychiatric history. Bereavement. Adaptation to bereavement will be measured using the Inventory of Complicated Grief (ICG).This is a 19 item self report measure of maladaptive symptoms of loss as described by the authors. Responses are given on a Likert scale.

PTSD. PTSD will be measured with both a clinician administered measure (CAPS) and a self-report measure (PDS).The CAPS is a 30 item interview that provides a diagnosis of PTSD based on all 17 symptoms of the DSM-IV defined disorder including frequency and intensity of symptoms. It also provides a measure of the impact of the symptoms on the patient's social and occupational functioning, the overall severity of the symptom complex, the patient's global improvement since baseline, and the validity of ratings obtained.

Depression. Depression will be measured with the SCID-I32 (described above) and the Beck Depression Inventory (BDI- II). The BDI (and subsequently, the BDI-II) is the most widely used instrument for measuring the severity of depression and a 'gold standard' among self-report measures of depression. It is a 21-item scale, with possible scores ranging from 0 to 63 (higher values correspond to higher depressive symptomatology).

Suicidality. Will be assessed with the Beck Scale for Suicide Assessment (BSS). This is a 21-item self-report instrument measuring the presence and severity of suicide ideation. Similar in format to the BDI, each item consists of three statements ranked in intensity from 0 to 2 Marital Impairment. The quality of adjustment in the marital relationship will be measured using the Dyadic Adjustment Scale (DAS). This 32 item measure is widely used in clinical and research settings and consists of four subscales: Dyadic Consensus, Dyadic Satisfaction, Dyadic Cohesion and Affectional Expression.

Social Impairment. Impairment in social functioning will be measured using the Social Adjustment Scale-Self Report which provides scores in the following domains: work, social and leisure activities, relations with extended family, primary relationship, parenthood, family life and economic.

Treatment Procedures. Referred persons will be screened and if they meet criteria will be matched as noted above for randomization. If persons do not meet criteria they will be referred for alternative treatment or to the community. Assessments will be conducted by our assessor/outreach coordinator. Each case will be reviewed at a consensus conference chaired by the PI.

Suicidal ideation and plans will be clinically assessed throughout the treatment protocol. Any participant identified at increased risk because of suicidal ideation will be monitored closely. A clinical consensus conference will be held and additional treatment will be recommended and provided as needed.

Treatment Fidelity. Treatment sessions will be audiotaped. Treatment fidelity raters will be trained to an 85% reliability level. Twenty-five percent of sessions will be randomly reviewed (stratifying for session number) and rated for adherence to protocol. Ten percent of sessions will be rated by a second rater to insure that reliability is maintained, guarding against rater drift.

DATA ANALYSES The design is a repeated measures (pre-treatment, post-treatment, 3 month follow-up) comparison of intervention and wait-list control conditions. We will assess treatment efficacy by examining the change from pre-treatment to the three-month follow-up score using an intent-to-treat analysis (carrying last observation forward). To avoid the loss of power associated with testing many hypotheses, we have selected a-priori as primary outcomes to be analyzed (1) complicated grief symptoms (ICG) and (2) marital adjustment. An analysis of change scores is equivalent to a repeated measures analysis comparing only baseline to three-month follow-up. For each outcome measure, an analysis of covariance using a change score will compare the intervention and wait-list conditions, controlling for the baseline score on the measure.

HUMAN SUBJECTS RESEARCH Sources of Data Baseline assessments will include demographic data, psychiatric history, current psychiatric diagnoses, description of the death of the child, relationship information, and social functioning information. Only staff working on the parental bereavement project will have access to subject identities. Any identifying subject data will be stored separately from the rest of the data. All data will be collected through in-person interviews and self-report questionnaires. All interviews will be videotaped for treatment adherence factors. This data will be collected specifically for this research project.

Potential Risks The principal risks for subjects participating in this study include possible emotional distress as they recall the painful story of the death of their child. The goal of the present clinical trial is to alleviate emotional distress on a long-term basis. It is also possible that subjects randomized to the wait-list control will have a deterioration of symptoms prior to participating in the research protocol. We will monitor this through weekly 15-minute phone check-ins to assess psychiatric status. Immediate treatment referral will be provided in the event of deterioration.

Recruitment and Informed Consent A referral system will be set-up through area churches and synagogues, parental bereavement support groups, different departments in Mt. Sinai Hospital (e.g. pediatrics, oncology, emergency medicine, etc), area funeral homes and Sloan Kettering Memorial Hospital. Members of the parent bereavement referral network will be provided with detailed descriptions of the program. Informed consent will be obtained in person after the research clinician presents a description of the treatment as well as the regulations regarding informed consent. They will be provided with written documentation of the above information. Ample time will be provided for potential subjects to ask questions. When it is clear that they understand the purpose of the study and the process of informed consent, they will be asked to sign and date the consent form if they agree to be in the study.

Protection of Subjects Well-Being While bereavement treatment research to date has shown no harm to subjects and some benefit, a system of monitoring the well being of participants will be put into place including the following procedures:

* All clinicians providing the manualized treatment will be licensed and trained in the techniques being applied.
* Prior to beginning the treatment protocol, intensive training and practice of the manualized treatment will be provided through formalized training sessions for all clinicians.
* Ongoing supervision will be provided throughout the duration of the treatment
* Patients randomized to the wait-list control will be monitored through weekly phone conversations.
* Referrals for any participants (focus groups, interviews, wait-list control study participants, family members involved in treatment) can be made for emergency or other inpatient or outpatient psychiatric services at Mt Sinai School of Medicine.

Protection of Data Any identifying subject data will be stored separately from all other patient data. While stored separately, both sets of data will be stored in a locked cabinet which will be in a locked room. Scientific presentations and publications will not use subject names and will only use aggregate data. Data entry will be done twice and compared to establish accuracy. After entry, data will be checked for variable ranges and internal consistency using SPSS.

Data and Safety Monitoring Plan A DSMB will be established to monitor the project. In addition, during all phases of the project, data collection will be monitored monthly by the PI through individual supervision, project team meetings and random review of session audiotapes and written transcripts. Monthly reports will be generated noting any problems encountered in treatment and the drop out of any participants. Any adverse events that occur during consent or treatment phases will be reported immediately to the PI. Adverse events will also be reported to the IRB and the NIH. Specifically, all serious adverse events associated with the study procedures, and/or any incidents involving the conduct of the study or patient participation, including problems with the consent processes will be reported. Summaries of safety and study performance information from reports will be provided to the IRB at the Mt. Sinai School of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Suffered the loss of a child between the ages of 0 and 25
* Loss occurred at least 6 months prior to beginning of study
* Score over 30 on the Inventory of Complicated Grief (ICG)
* Spouse living with identified patient and scoring less than 30 on the ICG

Exclusion Criteria:

* Parents under the age of 21
* Presence of overt psychosis as measured with the SCID
* Active substance abuse or dependence as measured with the SCID
* Suicidal or homicidal ideation as measured with the SCID and the BSS
* Suicidal or homicidal plans within the previous 6 months
* Initiation or change in psychotropic medication within the past 3 months
* Cognitive impairment precluding informed consent or ability to participate in treatment activities

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-01; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
complicated grief symptom change | change from pretreatment to 3 month follow-up
  Inventory of Complicated Grief

SECONDARY OUTCOMES:
marital adjustment change | change from pretreatment to 3 month follow-up
  Dyadic Adjustment Scale

CONTACTS AND LOCATIONS:
Overall Officials: Claude M Chemtob, Ph.D, Principal Investigator — Mount Sinai Medical School
Locations (1):
- The Israel Center for the Treatment of Psychotrauma, Jerusalem, Israel